CLINICAL TRIAL: NCT02394028
Title: A Phase III, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Etrolizumab as an Induction And Maintenance Treatment For Patients With Moderately to Severely Active Crohn's Disease
Brief Title: A Study to Assess Whether Etrolizumab is a Safe and Efficacious Treatment for Participants With Moderately to Severely Active Crohn's Disease
Acronym: BERGAMOT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA29144; 2014-003824-36 (EudraCT Number)
Record Dates: First submitted 2015-02-27; First posted 2015-03-20 (Estimated); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — etrolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg (Experimental): Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm will receive one subcutaneous (SC) injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
  Interventions: Drug: Etrolizumab; Drug: Placebo
- Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg (Experimental): Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm will receive one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
  Interventions: Drug: Etrolizumab; Drug: Placebo
- Induction Phase - Cohort 1 (Exploratory): Placebo (Placebo Comparator): Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm will receive two SC injections of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12 (and one SC injection of etrolizumab-matching placebo at Week 2) during the 14-week Induction Phase, in order to preserve the masking.
  Interventions: Drug: Placebo
- Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg (Experimental): Cohort 2 is enrolling participants after Cohort 1 and is considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm will receive one SC injection of open-label etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking for the dose of etrolizumab, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
  Interventions: Drug: Etrolizumab; Drug: Placebo
- Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg (Experimental): Cohort 2 is enrolling participants after Cohort 1 and is considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm will receive one SC injection of open-label etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking of the dose of etrolizumab, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
  Interventions: Drug: Etrolizumab; Drug: Placebo
- Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg (Experimental): Cohort 3 is the last to enroll participants (after Cohort 2) and will be the pivotal cohort for the Induction Phase. Participants randomized to this arm will receive one SC injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
  Interventions: Drug: Etrolizumab; Drug: Placebo
- Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg (Experimental): Cohort 3 is the last to enroll participants (after Cohort 2) and will be the pivotal cohort for the Induction Phase. Participants randomized to this arm will receive one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
  Interventions: Drug: Etrolizumab; Drug: Placebo
- Induction Phase - Cohort 3 (Pivotal): Placebo (Placebo Comparator): Cohort 3 is the last to enroll participants (after Cohort 2) and will be the pivotal cohort for the Induction Phase. Participants randomized to this arm will receive two SC injections of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12 (and one SC injection of etrolizumab-matching placebo at Week 2) during the 14-week Induction Phase, in order to preserve the masking.
  Interventions: Drug: Placebo
- Maintenance Phase - Placebo Responders: Placebo (Placebo Comparator): Participants who received placebo during the Induction Phase (from Cohorts 1 and 3) and achieved a CDAI-70 response at Week 14 will undergo a sham randomization into the Maintenance Phase. Placebo responders from induction will receive blinded maintenance treatment with an SC injection of placebo once every 4 weeks (q4w) from Week 16 to Week 64.
  Interventions: Drug: Placebo
- Maintenance Phase - Etrolizumab Responders: Placebo (Placebo Comparator): Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy will be re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm will receive blinded maintenance treatment with an SC injection of placebo q4w from Week 16 to Week 64.
  Interventions: Drug: Placebo
- Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg (Experimental): Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy will be re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm will receive blinded maintenance treatment with an SC injection of etrolizumab (105 mg) q4w from Week 16 to Week 64.
  Interventions: Drug: Etrolizumab

INTERVENTIONS:
Drug: Etrolizumab — Etrolizumab will be administered as per regimen specified in individual arms.
  Other Names: RO5490261; RG7413
  Arms: Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg; Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg; Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg; Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg; Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Drug: Placebo — Etrolizumab-matching placebo will be administered as per regimen specified in individual arms.
  Arms: Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg; Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg; Induction Phase - Cohort 1 (Exploratory): Placebo; Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg; Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg; Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Induction Phase - Cohort 3 (Pivotal): Placebo; Maintenance Phase - Etrolizumab Responders: Placebo; Maintenance Phase - Placebo Responders: Placebo

SUMMARY:
This is a multicenter, Phase 3, double-blind, placebo-controlled study evaluating the efficacy, safety, and tolerability of etrolizumab compared with placebo during induction and maintenance treatment of moderately to severely active Crohn's Disease (CD). The target population includes participants with CD who are refractory or intolerant to corticosteroids (CS) and/or immunosuppressant (IS) therapy and who have either not received prior anti-tumor necrosis factor (anti-TNF) therapy (TNF-naive) or who have had prior exposure to anti-TNF therapies and demonstrated inadequate responses or intolerance to anti-TNFs.

The study period will consist of a Screening Phase (up to 35 days) plus (+) a 14-week Induction Phase + a 52-week Maintenance Phase + a 12-week Safety Follow-up Phase. At Week 14 (end of Induction Phase), participants achieving a decrease from baseline of at least 70 points in the Crohn's Disease Activity Index (CDAI) score (CDAI-70 response) without the use of rescue therapy will continue to the Maintenance Phase.

ELIGIBILITY:
Inclusion Criteria:

* Moderately to severely active Crohn's Disease (CD) as determined by the CDAI, patient reported outcomes and endoscopically defined disease activity in the ileum and/or colon
* Intolerance, refractory disease, or no response to corticosteroids (CS), immunosuppressants (IS), or anti-TNF therapy within 5 years from screening. Participants who have not previously demonstrated inadequate response or intolerance to one or more anti-TNF therapies are eligible to participate in the study provided they are intolerant or refractory to CS or IS therapy
* Use of effective contraception as defined by the protocol

Exclusion Criteria:

* A history of, or current conditions affecting the digestive tract, such as ulcerative colitis, indeterminate colitis, fistulizing disease, abdominal or perianal abscess, adenomatous colonic polyps not excised, colonic mucosal dysplasia, and short bowel syndrome
* Planned surgery for CD
* Ileostomy or colostomy
* Has received non-permitted inflammatory bowel disease (IBD) therapies (including natalizumab, vedolizumab, and efalizumab, as stated in the protocol)
* Any prior treatment with ustekinumab within 14 weeks prior to randomization
* Chronic hepatitis B or C infection, human immunodeficiency virus (HIV), active or latent tuberculosis (participants with prior history of Bacillus Calmette-Guérin [BCG] vaccination must pass protocol-defined screening criteria)
* Sinus tract with evidence for infection (e.g., purulent discharge) in the clinical judgment of the investigator. Fistulas related to CD are not exclusionary
* Any prior treatment with anti-adhesion molecules (e.g., anti-mucosal addressin cell adhesion molecule [anti-MAdCAM-1])
* Any major episode of infection requiring treatment with intravenous antibiotics ≤8 weeks prior to screening or oral antibiotics ≤4 weeks prior to screening. Treatment with antibiotics as adjunctive therapy for CD in the absence of documented infection is not exclusionary
* Hospitalization (other than for elective reasons) within 4 weeks prior to randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2015-03-20 (Actual); Primary Completion 2021-09-07 (Actual); Study Completion 2021-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (327):
- United States (62):
  - Valley Gastroenterology Consultants, Arcadia, California
  - University of California San Diego Medical Center, La Jolla, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Digestive Care Associates, A Medical Corporation, San Carlos, California
  - SDG Clinical Research, San Diego, California
  - University of California at San Francisco (PARENT); Gastroenterology, Hepatology & Nutrition, San Francisco, California
  - Peak Gastroenterology Associates; Gastroenterology, Colorado Springs, Colorado
  - Innovative Medical Research of South Florida, Aventura, Florida
  - West Central Gastroenterology d/b/a Gastro Florida, Clearwater, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - IMIC, Inc, Miami Beach, Florida
  - FQL Research, LLC, Miramar, Florida
  - Advanced Research Institute, Inc., Trinity, Florida
  - Shafran Gastroenterology Center, Winter Park, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Atlanta, Georgia
  - Gastrointestinal Diseases Research, Columbus, Georgia
  - Atlanta Center for Gastroenterology, PC, Decatur, Georgia
  - Gastroenterology Associates of Central Georgia, Macon, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Advanced Clinical Research, Meridian, Idaho
  - Northwestern University-Feinberg School of Medicine; Division of Gastroenterology and Hepatology, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - Southwest Gastroenterology; DM Clinical Research, Oak Lawn, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Gastroenterology Associates, LLC, Baton Rouge, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Gastroenterology Associates of Western Michigan, P.L.C., Grand Rapids, Michigan
  - Center for Digestive Health, Troy, Michigan
  - Henry Ford Health System, West Bloomfield, Michigan
  - Mayo Clinic - Rochester; Gastrology, Rochester, Minnesota
  - University of Mississippi Medical Center; Division of Gastroenterology, Jackson, Mississippi
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Concorde Medical Group, New York, New York
  - Weill Cornell Medical College (WCMC) - Judith Jaffe Multiple Sclerosis Center (JJMSC), New York, New York
  - Lenox Hill Hospital, New York, New York
  - University of North Carolina At Chapel Hill, Chapel Hill, North Carolina
  - Charlotte Gastroenterology and Hepatology, P.L.L.C, Charlotte, North Carolina
  - Kinston Medical Specialists, Kinston, North Carolina
  - Consultants for Clinical Research Inc., Cincinnati, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Digestive Disease Specialists, Inc., Oklahoma City, Oklahoma
  - Great Lakes Medical Research, LLC, Harrisburg, Pennsylvania
  - Innovative Clinical Research, Greenville, South Carolina
  - Gastroenterology Center of the MidSouth PC, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Digestive Disease Consultants - Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center; Internal Medicne, Dallas, Texas
  - Baylor College of Medicine; Gastroenterology, Houston, Texas
  - Methodist Hospital Research Institute, Houston, Texas
  - Wellness Clinical Research Center, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Ericksen Research and Development, Clinton, Utah
  - University of Utah School of Medicine, Salt Lake City, Utah
  - McGuire Research Institute; Gastroenterology, Richmond, Virginia
  - Digestive Disease Institute; Virginia Mason Medical Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Hospital Italiano, Buenos Aires, Argentina
- Australia (15):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Bankstown-Lidcombe Hospital, Bankstown, New South Wales
  - Concord Repatriation General Hospital, Concord, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - University of the Sunshine Coast, Sippy Downs, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Bedford Park, South Australia
  - Monash Medical Centre Clayton, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Footscray Hospital; Gastroenterology, Footscray, Victoria
  - St Frances Xavier Cabrini Hospital, Malvern, Victoria
  - Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital; Department of Colorectal Medicine and Genetics, Parkville, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (2):
  - LKH - Universitätsklinikum der PMU Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (5):
  - CHU St Pierre (St Pierre), Brussels
  - Hospital Erasme, Brussels
  - UZ Brussel, Brussels
  - UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
- Brazil (17):
  - L2IP -Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - Instituto Goiano de Gastroenterologia e Endoscopia Digestiva Ltda, Goiânia, Goiás
  - Hospital Felicio Rocho, Belo Horizonte, Minas Gerais
  - Centro Digestivo de Curitiba, Curitiba, Paraná
  - Hospital Universitario Clementino Fraga Filho - UFRJ; Gastroenterologia, Rio de Janeiro, Rio de Janeiro
  - Instituto Brasil de Pesquisa Clínica-IBPCLIN S/A, Rio de Janeiro, Rio de Janeiro
  - Hospital São Vicente de Paulo; Institute of Education and Reseach / Cardiovascular Research Unit, Passo Fundo, Rio Grande do Sul
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital Ernesto Dornelles, Porto Alegre, Rio Grande do Sul
  - UNESP - Faculdade de Medicina da Universidade Estadual Paulista - Campus Botucatu, Botucatu, São Paulo
  - Pesquisare Saúde Sociedade Simples, Santo André, São Paulo
  - Praxis Pesquisa Médica, Santo André, São Paulo
  - Hospital Estadual Mario Covas, Santo André, São Paulo
  - Hospital de Base de Sao Jose do Rio Preto, São José do Rio Preto, São Paulo
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Hospital Sao Paulo, São Paulo, São Paulo
  - Hospital do Servidor Público Estadual/HSPE-SP, São Paulo, São Paulo
- Bulgaria (3):
  - "City Clinic UMHAC" EOOD, Sofia
  - UMHAT "Sv. Ivan Rilski", EAD, Sofia
  - UMHAT Tsaritsa Yoanna - ISUL, EAD, Sofia
- Canada (13):
  - University of Calgary, Calgary, Alberta
  - Zeidler Ledcor Centre - University of Alberta; Division of Gasroenterology, Edmonton, Alberta
  - (G.I.R.I.) GI Research Institute, Vancouver, British Columbia
  - Winnipeg Regional Health Authority, Winnipeg, Manitoba
  - Queen Elizabeth II Health Sciences Centre; Gastroenterology Research, Halifax, Nova Scotia
  - University Hospital - London Health Sciences Centre, London, Ontario
  - Taunton Health Centre, Oshawa, Ontario
  - The Ottawa Hospital - Riverside Campus; Gastrointestinal Clinical Research Unit, Ottawa, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Toronto Digestive Disease Associates, Vaughan, Ontario
  - Hôpital Maisonneuve - Rosemont, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - Royal University Hospital, Saskatoon, Saskatchewan
- Croatia (4):
  - Clinical Hospital Centre Osijek, Osijek
  - General Hospital Pula, Pula
  - Clinical Hospital Center Sestre Milosrdnice, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (10):
  - Vojenska nemocnice Brno, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - Nemocnice Ceske Budejovice a.s., České Budějovice
  - Gastroenterologie s.r.o., Hradec Králové
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - PreventaMed, s.r.o., Olomouc
  - Fakultni nemocnice Ostrava, Ostrava - Poruba
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Klinicke centrum ISCARE Lighthouse, Prague
- Estonia (3):
  - West Tallinn Central Hospital, Tallinn
  - North Estonia Medical Centre Foundation, Tallinn
  - Tartu University Hospital, Tartu
- France (14):
  - CHU Amiens - Hopital Sud, Amiens
  - CHU de Caen - Hopital Cote de Nacre, Caen
  - Hôpital Beaujon, Clichy
  - Hopital Claude Huriez - CHU Lille, Lille
  - CHU NANTES - Hôtel Dieu; Pharmacy, Nantes
  - CHU Nice - Hopital de l'Archet 2, Nice
  - Hôpital Saint-Louis, Paris
  - Groupe Hospitalier Sud - Hôpital Haut-Lévêque - USN, Pessac
  - Centre Hospitalier Lyon Sud; Service de Gastro-Enterologie, Pierre-Bénite
  - CHU du Reims - Hopital Robert Debré, Reims
  - CHU Rennes - Hopital Pontchaillou, Rennes
  - CHU Saint Etienne - Hôpital Nord, Saint-Etienne
  - Höpital Hautepierre; Pediatrie1, Strasbourg
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy
- Germany (11):
  - Charite-Campus Virchow Klinikum; Hepatologie und Gastroenterologie, Berlin
  - Krankenhaus Waldfriede e. V., Berlin
  - Berufsgenossenschaftliches Universitaetsklinikum Bergmannsheil GmbH, Bochum
  - Universitätsklinikum Koeln, Cologne
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt
  - Universitaetsklinikum Halle (Saale), Halle
  - Medizinische Hochschule Hannover; Gastroenterology and Hepatology dept, Hanover
  - Klinikum Mannheim GmbH Universitätsklinikum, Mannheim
  - Gemeinschaftspraxis, Offenburg
  - Universitaetsklinikum Tuebingen, Tübingen
  - Universitaetsklinikum Ulm, Ulm
- Hungary (10):
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaza, Békéscsaba
  - Obudai Egeszsegugyi Centrum Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Eszak-Kozep-budai Centrum, Uj Szent Janos Korhaz es Szakrendelo, Budapest
  - Pannonia Maganorvosi Centrum, Budapest
  - Debreceni Egyetem, Debrecen
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Pest Megyei Flor Ferenc Korhaz, Kistarcsa
  - Pecsi Tudomanyegyetem, Pécs
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
- Israel (8):
  - Haemek Medical Center, Afula
  - Soroka University Medical Centre, Beersheba
  - Wolfson Medical Center; Obstetrics and Gynecology, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Holy Family Hospital, Nazareth
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Tel Aviv Sourasky Medical Center; Pharmacy, Tel Aviv
- Italy (10):
  - A.O.U. Policlinico di Modena, Modena, Emilia-Romagna
  - Azienda Ospedaliera San Camillo Forlanini, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli; Farmacia, Rome, Lazio
  - Asst Fatebenefratelli Sacco (Fatebenefratelli), Milan, Lombardy
  - ASST FATEBENEFRATELLI SACCO (Sacco), Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Niguarda (Grande Ospedale Metropolitano Niguarda), Milan, Lombardy
  - Istituto Clinico Humanitas, Rozzano (MI), Lombardy
  - I.R.C.C.S Policlinico San Donato, San Donato Milanese (MI), Lombardy
  - Ospedale Umberto I di Torino, Turin, Piedmont
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
- Latvia (2):
  - Riga East Clinical University Hospital; Clinic Gailezers, Riga
  - Pauls Stradins Clinical University Hospital, Riga
- Lithuania (2):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Vilnius University Hospital Santariskiu Clinic, Public Institution; Cardiology, Vilnius
- Mexico (2):
  - Clinical Research Institute, Tlalnepantla, Mexico CITY (federal District)
  - Medical Care & Research SA de CV, Mérida, Yucatán
- Netherlands (7):
  - Amsterdam UMC, Locatie VUMC; Neurology, Amsterdam
  - Amsterdam UMC Location AMC, Amsterdam
  - Leids Universitair Medisch Centrum, Leiden
  - Maastricht University Medical Center, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - Zuyderland Medisch Centrum - Sittard Geleen, Sittard-Geleen
  - ETZ TweeSteden, Tilburg
- New Zealand (6):
  - North Shore Hospital, Auckland
  - Christchurch Hospital NZ, Christchurch
  - Dunedin Public Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Shakespeare Specialist Group, Takapuna
  - Tauranga Hospital, Tauranga
- Poland (19):
  - SP ZOZ Wojewodzki Szpital Zespolony im. J. Sniadeckiego, Bialystok
  - Nasz Lekarz Osrodek Badan Klinicznych, Bydgoszcz
  - Elblaski Szpital Specjalistyczny z Przychodnia SP ZOZ, Elblag
  - ETG Kielce, Kielce
  - Centrum Opieki Zdrowotnej Orkan-Med, Ksawerów
  - Indywidualna Specjalistyczna Praktyka Lekarska, Lublin
  - Allmedica Badania Kliniczne Sp z o.o. Sp K., Nowy Targ
  - Centrum Medyczne "MEDYK", Rzeszów
  - Gabinet Lekarski, Bartosz Korczowski, Rzeszów
  - Specjalistyczna Praktyka Lekarska Dr med. Marek Horynski; endoskopia, Sopot
  - Niepubliczny Zaklad Opieki Zdrowotnej SONOMED, Szczecin
  - Twoja Przychodnia-Szczecinskie Centrum Medyczne, Szczecin
  - Gastromed Kopon Zmudzinski i Wspolnicy Sp.j.Specjalistyczne Centrum Gastrologii i Endoskopii Specj, Torun
  - Centrum Zdrowia MDM, Warsaw
  - Warsaw IBD Point Profesor Kierkus, Warsaw
  - Zespó Przychodni Specjalistycznych PRIMA, Warsaw
  - PlanetMed sp. z o.o., Wroclaw
  - LexMedica Osrodek Badan Klinicznych, Wroclaw
  - EuroMediCare Szpital Specjalistyczny z Przychodnią we Wrocławiu, Wroclaw
- Romania (3):
  - S.C MedLife S.A, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Centrul de Gastroenterologie Dr. Goldis, Timișoara
- Russia (12):
  - Yusupov Hospital, Moskva, Adygeya Republic
  - LLC "Novosibirsk GastroCenter", Novosibirsk, Altaj
  - North-Western Medical University n.a. I.I. Mechnikov; Rheumatology, Saint Petersburg, Sankt-Peterburg
  - Baltic Medicine, Saint Petersburg, Sankt-Peterburg
  - SBIH City Clinical Hospital #31, Saint Petersburg, Sankt-Peterburg
  - SBEI HPE Altai StateMedicalUniversityofMoH andSD, Barnaul
  - Irkutsk State Medical Academy of Continuing Education, Irkutsk
  - SBEIHPE Novosibirsk State Medical University, Novosibirsk
  - BHI of Omsk region Clinical Oncology Dispensary, Omsk
  - Evromedservis LCC, Pushkin
  - SEIHPE "Rostov SMU of MoH of RF", Rostov-on-Don
  - Federal State Military Educational Institution; High Professional Education Military Medical Acad, Saint Petersburg
- Serbia (5):
  - Clinical Helth Centre Zvezdara, Belgrade
  - Military Medical Academy, Belgrade
  - University Hospital Medical Center Bezanijska kosa, Belgrade
  - Clinical Center of Vojvodina, Novi Sad
  - General Hospital Djordje Joanovic, Zrenjanin
- Slovakia (4):
  - IBDcentrum s.r.o., Bratislava
  - KM Management spol. s r.o., Nitra
  - Accout Center s.r.o., Šahy
  - Endomed, s.r.o., Vranov nad Topľou
- South Africa (2):
  - Dr D Epstein Practice, Cape Town
  - Emmed Research, Pretoria
- South Korea (15):
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kyungpook National University Hospital, Daegu
  - Yeungnam Univ. Hospital, Daegu
  - Hanyang University Guri Hospital, Gyeonggi-do
  - Korea University Ansan Hospital, Gyeonggi-do
  - CHA Bundang Medical Centre; CHA university, Seongnam
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Yonsei University Wonju Severance Christian Hospital, Wŏnju
- Spain (14):
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario Puerta de Hierro Majadahonda; Hepatology studies, Majadahonda, Madrid
  - Hospital Clínic i Provincial; Servicio de Farmacia, Barcelona
  - Centro Médico Teknon, Barcelona
  - Hospital Reina Sofia; Medical Oncology, Córdoba
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital Universitario de la Princesa, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Complejo Hospitalario de Pontevedra, Pontevedra
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (3):
  - Inselspital-Universitaetsspital Bern, Bern
  - Crohn-Colitis Zentrum Bern - Gemeinschaftspraxis Balsiger, Seibold und Partner, Bern
  - Universitätsspital Zürich, Zurich
- Turkey (Türkiye) (9):
  - Ankara University Medical Faculty, Ankara
  - Hacettepe University Medical Faculty; Gastroenterology, Ankara
  - Gazi University Medical Faculty, Ankara
  - Acibadem Fulya Hospital; Neurology, Istanbul
  - Haydarpasa Numune Training and Research Hospital; Medical Oncology, Istanbul
  - Medeniyet University Goztepe Training and Research Hospital; Chest Diseases, Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli Universitesi Tip Fakultesi; Infectious Diseases, Kocaeli
  - Acibadem Kozyatagi Hospital; Gastroenterology, Kozyataği
- Ukraine (19):
  - CHI Prof.O.O.Shalimov Kharkiv City Clinical Hospital #2, Kharkiv, Kharkiv Governorate
  - CI of Healthcare Kharkiv Reg Clin Hosp-Center of Med Emergency & Accident Medicine, Kharkiv, Kharkiv Governorate
  - Medical Center of Limited Liability Company Medical Clinic Blagomed, Kyiv, KIEV Governorate
  - Med Center of International Institute of Clinical Trials LLC; Medical Center "OK!Clinic+", Kyiv, KIEV Governorate
  - CI of Kyiv RC Regional Clinical Hospital #2, Kyiv, KIEV Governorate
  - Lviv Regional Clinical Hospital, Lviv, KIEV Governorate
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk, Kuban People's Republica
  - RCNECRCH Dept of Surgery, SHEI Ukr BSMU, Chernivtsi, Podolia Governorate
  - Kremenchuk first city hospital n.a. O.T. Bohaievskyi; Gastroenterology department, Kremenchuk, Poltava Governorate
  - CI City Hospital #1, Zaporizhzhia, Tavria Okruha
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - CHI Kharkiv City Clinical Hospital #13, Kharkiv
  - Kyiv CCH #18 Dept of Proctology O. O. Bogomolets NMU, Kyiv
  - City Hospital #1, Mykolaiv
  - Railway Transport Odesa CH of Healthcare Ctr Branch of PJSC Ukrainian Railway Dept of Therapy #2, Odesa
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - M.I. Pyrogov VRCH Dept of Gastroenterology M.I. Pyrogov VNMU, Vinnytsia
  - MCIC MC LLC Health Clinic, Vinnytsia
  - LLC Diaservis, Zaporizhzhia
- United Kingdom (15):
  - Royal Victoria Hospital, Belfast
  - Addenbrooke's Hospital, Cambridge
  - University Hospital Coventry, Coventry
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Queen Elizabeth Hospital, Kings Lynn
  - St James University Hospital, Leeds
  - Royal Liverpool University Hospital, Liverpool
  - Whipps Cross Hospital, London
  - University College London Hospital, London
  - Fairfield General Hospital, Manchester
  - Royal Victoria Infirmary; Stroke unit, Newcastle upon Tyne
  - Nottingham University Hospitals Queen's Medical Centre, Nottingham
  - Royal Berkshire Hospital, Reading
  - Southampton General Hospital, Southampton
  - Royal Wolverhampton hospital; McHale Building, Wolverhampton

REFERENCES:
- [Derived] Sandborn WJ, Panes J, Danese S, Sharafali Z, Hassanali A, Jacob-Moffatt R, Eden C, Daperno M, Valentine JF, Laharie D, Baia C, Atreya R, Panaccione R, Rydzewska G, Aguilar H, Vermeire S; BERGAMOT Study Group. Etrolizumab as induction and maintenance therapy in patients with moderately to severely active Crohn's disease (BERGAMOT): a randomised, placebo-controlled, double-blind, phase 3 trial. Lancet Gastroenterol Hepatol. 2023 Jan;8(1):43-55. doi: 10.1016/S2468-1253(22)00303-X. Epub 2022 Oct 12. PMID 36240801
- [Derived] Dai B, Hackney JA, Ichikawa R, Nguyen A, Elstrott J, Orozco LD, Sun KH, Modrusan Z, Gogineni A, Scherl A, Gubatan J, Habtezion A, Deswal M, Somsouk M, Faubion WA, Chai A, Sharafali Z, Hassanali A, Oh YS, Tole S, McBride J, Keir ME, Yi T. Dual targeting of lymphocyte homing and retention through alpha4beta7 and alphaEbeta7 inhibition in inflammatory bowel disease. Cell Rep Med. 2021 Aug 17;2(8):100381. doi: 10.1016/j.xcrm.2021.100381. eCollection 2021 Aug 17. PMID 34467254
- [Derived] Reinisch W, Mishkin DS, Oh YS, Schreiber S, Hussain F, Jacob R, Hassanali A, Daperno M. Impact of various central endoscopy reading models on treatment outcome in Crohn's disease using data from the randomized, controlled, exploratory cohort arm of the BERGAMOT trial. Gastrointest Endosc. 2021 Jan;93(1):174-182.e2. doi: 10.1016/j.gie.2020.05.020. Epub 2020 May 25. PMID 32464142
- [Derived] Sandborn WJ, Vermeire S, Tyrrell H, Hassanali A, Lacey S, Tole S, Tatro AR; Etrolizumab Global Steering Committee. Etrolizumab for the Treatment of Ulcerative Colitis and Crohn's Disease: An Overview of the Phase 3 Clinical Program. Adv Ther. 2020 Jul;37(7):3417-3431. doi: 10.1007/s12325-020-01366-2. Epub 2020 May 22. PMID 32445184

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At the time of study closure, a total of 1035 patients were randomized into the induction phase, enrolled sequentially across Cohorts 1, 2, and 3. The final sample size for the pivotal induction Cohort 3 was lower than the 496 patients planned per the final protocol due to the early closure of the study. Cohorts below are mutually exclusive.
Pre-assignment Details: A total of 1035 participants entered the study across induction cohorts 1-3, a subset of 487 patients moved into the maintenance phase of the study.
Groups:
- Placebo Cohort 1: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received two SC injections of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12 (and one SC injection of etrolizumab-matching placebo at Week 2) during the 14-week Induction Phase, in order to preserve the masking.
- Etrolizumab 105mg Cohort 1: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Etrolizumab 210mg Cohort 1: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one SC injection of etrolizumab (210 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Etrolizumab 105mg Cohort 2: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking of the dose of etrolizumab, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Etrolizumab 210mg Cohort 2: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (210 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking of the dose of etrolizumab, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Placebo Cohort 3: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received two SC injections of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12 (and one SC injection of etrolizumab-matching placebo at Week 2) during the 14-week Induction Phase, in order to preserve the masking.
- Etrolizumab 105mg Cohort 3: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Etrolizumab 210mg Cohort 3: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Placebo/Placebo: Participants who received placebo during the Induction Phase (from Cohorts 1 and 3) and achieved a CDAI-70 response at Week 14 underwent a sham randomization into the Maintenance Phase. Placebo responders from induction received blinded maintenance treatment with an SC injection of placebo once every 4 weeks (q4w) from Week 16 to Week 64.
- Etrolizumab/Placebo: Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who were re-randomized to this arm received blinded maintenance treatment with an SC injection of placebo q4w from Week 16 to Week 64.
- Etrolizumab/Etrolizumab 105mg: Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who were re-randomized to this arm received blinded maintenance treatment with an SC injection of etrolizumab (105 mg) q4w from Week 16 to Week 64.
Period: Induction Phase
Arm/Group | Placebo Cohort 1 | Etrolizumab 105mg Cohort 1 | Etrolizumab 210mg Cohort 1 | Etrolizumab 105mg Cohort 2 | Etrolizumab 210mg Cohort 2 | Placebo Cohort 3 | Etrolizumab 105mg Cohort 3 | Etrolizumab 210mg Cohort 3 | Placebo/Placebo | Etrolizumab/Placebo | Etrolizumab/Etrolizumab 105mg
Started | 59 | 120 | 121 | 176 | 174 | 97 | 143 | 145 | 0 | 0 | 0
Completed | 52 | 104 | 108 | 141 | 145 | 80 | 118 | 114 | 0 | 0 | 0
Not Completed | 7 | 16 | 13 | 35 | 29 | 17 | 25 | 31 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 4 | 1 | 2 | 5 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 6 | 2 | 17 | 14 | 8 | 17 | 23 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Non-compliance | 0 | 1 | 3 | 1 | 3 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 4 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 2 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 4 | 6 | 7 | 4 | 3 | 6 | 0 | 0 | 0
Not completed — Early withdrawal and roll over to a different study | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Sponsor decision | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Technical reason | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — :ack of calculation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Maintenance Phase
Arm/Group | Placebo Cohort 1 | Etrolizumab 105mg Cohort 1 | Etrolizumab 210mg Cohort 1 | Etrolizumab 105mg Cohort 2 | Etrolizumab 210mg Cohort 2 | Placebo Cohort 3 | Etrolizumab 105mg Cohort 3 | Etrolizumab 210mg Cohort 3 | Placebo/Placebo | Etrolizumab/Placebo | Etrolizumab/Etrolizumab 105mg
Started | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 0 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive either placebo or etrolizumab 105 mg.) | 53 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive placebo.) | 217 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive placebo.) | 217 (Participants from the induction phase who had achieved a CDAI-70 response without the use of rescue therapy were enrolled in the maintenance phase to receive etrolizumab 105 mg.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 41 | 175 | 165
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12 | 42 | 52
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 2
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7 | 25 | 33
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Site closure | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 12 | 12

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants randomized who received at least one dose of study treatment, grouped under the treatment arm received.
Groups:
- Maintenance Phase - Placebo Responders: Placebo: Participants who received placebo during the Induction Phase (from Cohorts 1 and 3) and achieved a CDAI-70 response at Week 14 underwent a sham randomization into the Maintenance Phase. Placebo responders from induction received blinded maintenance treatment with an SC injection of placebo once every 4 weeks (q4w) from Week 16 to Week 64.
- Maintenance Phase - Etrolizumab Responders: Placebo: Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm received blinded maintenance treatment with an SC injection of placebo q4w from Week 16 to Week 64.
- Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg: Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm received blinded maintenance treatment with an SC injection of etrolizumab (105 mg) q4w from Week 16 to Week 64.
- Total: Total of all reporting groups
Arm/Group | Placebo Cohort 1 | Etrolizumab 105mg Cohort 1 | Etrolizumab 210mg Cohort 1 | Etrolizumab 105mg Cohort 2 | Etrolizumab 210mg Cohort 2 | Placebo Cohort 3 | Etrolizumab 105mg Cohort 3 | Etrolizumab 210mg Cohort 3 | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg | Total
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217 | 1521
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Induction Phase: Number analyzed is for participants in induction phase.
  Maintenance Phase: Number analyzed is for participants who entered the maintenance phase
  Years
    Induction Phase: number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0 | 1034
    Induction Phase | 36.5 (12.7) | 38.9 (13.1) | 38.6 (13.4) | 38.4 (13.3) | 38.2 (13.2) | 37.1 (13.6) | 38.3 (13.4) | 36.5 (13.1) |  |  |  | 37.9 (13.2)
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 217 | 217 | 487
    Maintenance Phase |  |  |  |  |  |  |  |  | 38.2 (13.3) | 37.9 (12.6) | 38.8 (12.9) | 38.3 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Induction Phase: Number analyzed is for participants in induction phase. Maintenance Phase: Number analyzed is for participants who entered the maintenance phase.
  Participants
    Induction Phase: number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0 | 1034
    Induction Phase: Female | 31 | 57 | 68 | 80 | 80 | 38 | 69 | 69 |  |  |  | 492
    Induction Phase: Male | 28 | 63 | 53 | 96 | 94 | 58 | 74 | 76 |  |  |  | 542
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 217 | 217 | 487
    Maintenance Phase: Female |  |  |  |  |  |  |  |  | 24 | 118 | 98 | 240
    Maintenance Phase: Male |  |  |  |  |  |  |  |  | 29 | 99 | 119 | 247
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Induction Phase: Number analyzed is for participants in induction phase. Maintenance Phase: Number analyzed is for participants who entered the maintenance phase.
  Participants
    Induction Phase: number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0 | 1034
    Induction Phase: Hispanic or Latino | 2 | 5 | 5 | 7 | 8 | 15 | 13 | 7 |  |  |  | 62
    Induction Phase: Not Hispanic or Latino | 53 | 110 | 113 | 160 | 154 | 74 | 126 | 129 |  |  |  | 919
    Induction Phase: Unknown or Not Reported | 4 | 5 | 3 | 9 | 12 | 7 | 4 | 9 |  |  |  | 53
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 217 | 217 | 487
    Maintenance Phase: Hispanic or Latino |  |  |  |  |  |  |  |  | 7 | 10 | 12 | 29
    Maintenance Phase: Not Hispanic or Latino |  |  |  |  |  |  |  |  | 41 | 199 | 197 | 437
    Maintenance Phase: Unknown or Not Reported |  |  |  |  |  |  |  |  | 5 | 8 | 8 | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — race Population: Induction Phase: Number analyzed is for participants in induction phase. Maintenance Phase: Number analyzed is for participants who entered the maintenance phase.
  Participants
    Induction Phase: number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0 | 1034
    Induction Phase: American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 |  |  |  | 4
    Induction Phase: Asian | 5 | 9 | 7 | 8 | 14 | 0 | 4 | 2 |  |  |  | 49
    Induction Phase: Black or African American | 3 | 5 | 2 | 1 | 5 | 6 | 8 | 2 |  |  |  | 32
    Induction Phase: White | 46 | 96 | 104 | 153 | 141 | 80 | 117 | 128 |  |  |  | 865
    Induction Phase: Other | 1 | 2 | 2 | 4 | 2 | 3 | 3 | 5 |  |  |  | 22
    Induction Phase: Multiple | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 |  |  |  | 3
    Induction Phase: Unknown | 4 | 7 | 5 | 10 | 12 | 6 | 8 | 7 |  |  |  | 59
    Maintenance Phase: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 53 | 217 | 217 | 487
    Maintenance Phase: American Indian or Alaska Native |  |  |  |  |  |  |  |  | 1 | 0 | 0 | 1
    Maintenance Phase: Asian |  |  |  |  |  |  |  |  | 0 | 8 | 11 | 19
    Maintenance Phase: Black or African American |  |  |  |  |  |  |  |  | 2 | 5 | 9 | 16
    Maintenance Phase: White |  |  |  |  |  |  |  |  | 45 | 193 | 182 | 420
    Maintenance Phase: Other |  |  |  |  |  |  |  |  | 2 | 4 | 7 | 13
    Maintenance Phase: Multiple |  |  |  |  |  |  |  |  | 0 | 1 | 1 | 2
    Maintenance Phase: Unknown |  |  |  |  |  |  |  |  | 3 | 6 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Induction Phase: Cohort 1: Percentage of Participants With Clinical Remission at Week 14
Description: Clinical remission is defined as liquid/soft stool frequency (SF) mean daily score less than or equal (≤)3 and abdominal pain mean daily score ≤1, with no worsening in either subscore compared to baseline, averaged over the 7 days prior to visit.
Time Frame: Week 14
Population: mITT - Modified Intent to Treat population: all patients randomized who received at least one dose of study drug, grouped under the randomized treatment arm. Results for Induction Phase Cohort 2 and 3 and Maintenance Phase are not presented.
Measure: Number (90% Confidence Interval); unit: Percentage of Particiapnts
Groups:
- Induction Phase - Cohort 1 (Exploratory): Placebo: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received two SC injections of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12 (and one SC injection of etrolizumab-matching placebo at Week 2) during the 14-week Induction Phase, in order to preserve the masking. 90%CI
- Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12. 90%CI
- Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one subcutaneous (SC) injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12. 90%CI
- Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking of the dose of etrolizumab, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking for the dose of etrolizumab, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Induction Phase - Cohort 3 (Pivotal): Placebo: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received two SC injections of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12 (and one SC injection of etrolizumab-matching placebo at Week 2) during the 14-week Induction Phase, in order to preserve the masking.
- Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of Particiapnts | 11.9 [6.56 to 20.51] | 20.00 [14.69 to 26.64] | 27.3 [21.16 to 34.37] |  |  |  |  |  |  |  |

2. Primary Outcome: Induction Phase: Cohort 2 and 3: Percentage of Participants With Clinical Remission at Week 14
Description: as for outcome 1
Time Frame: Week 14
Population: mITT - Modified Intent to Treat population: all patients randomized who received at least one dose of study drug, grouped under the randomized treatment arm. Results for Induction Phase Cohort 1 and Maintenance Phase are not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Particiapnts
Groups:
- Induction Phase - Cohort 1 (Exploratory): Placebo: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received two SC injections of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12 (and one SC injection of etrolizumab-matching placebo at Week 2) during the 14-week Induction Phase, in order to preserve the masking.
- Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one subcutaneous (SC) injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0
Percentage of Particiapnts |  |  |  | 29.5 [23.30 to 36.66] | 29.3 [23.05 to 36.46] | 29.2 [21.02 to 38.92] | 30.1 [23.16 to 38.03] | 33.1 [25.97 to 41.11] |  |  |
Statistical Analysis 1: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Test type: Superiority; p = 0.8508, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 1.1, 95% CI 2-sided [-10.85 to 12.56] — Difference in remission rates is adjusted using CMH weights and the 95% CIs use the Newcombes method
Statistical Analysis 2: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Test type: Superiority; p = 0.5235, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 3.8, 95% CI 2-sided [-8.30 to 15.27] — Difference in remission rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

3. Primary Outcome: Induction Phase: Cohort 1: Percentage of Participants With Endoscopic Improvement at Week 14
Description: Endoscopic improvement is defined as 50 percent (%) reduction from baseline in Simplified Endoscopic Index for Crohn's Disease (SES-CD) score.
Time Frame: Week 14
Population: mITT. Results for Induction Phase Cohort 2 and 3 and Maintenance Phase are not presented.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking for the dose of etrolizumab, participants will also receive one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 3.4 [-1.74 to 8.52] | 19.5 [12.37 to 26.64] | 16.8 [10.11 to 23.50] |  |  |  |  |  |  |  |

4. Primary Outcome: Induction Phase: Cohort 2 and 3: Percentage of Participants With Endoscopic Improvement at Week 14
Description: as for outcome 3
Time Frame: Week 14
Population: mITT. Results for Induction Phase Cohort 1 and Maintenance Phase are not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0
Percentage of Participants |  |  |  | 20.8 [14.81 to 26.86] | 22.2 [16.02 to 28.35] | 21.6 [13.24 to 29.95] | 26.2 [18.96 to 33.44] | 27.4 [20.01 to 34.79] |  |  |
Statistical Analysis 1: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Test type: Superiority; p = 0.7908, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 4.9, 95% CI 2-sided [-6.26 to 16.11] — Difference in response rates is adjusted using CMH weights and the 95% CIs use the Newcombes method
Statistical Analysis 2: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Test type: Superiority; p = 0.3170, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 5.8, 95% CI 2-sided [-5.43 to 17.05] — Difference in response rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

5. Primary Outcome: Maintenance Phase: Percentage of Participants With Clinical Remission at Week 66
Description: Clinical remission is defined as SF mean daily score ≤3 and abdominal pain mean daily score ≤1, with no worsening in either subscore compared to baseline, averaged over the 7 days prior to visit.
  Maintenance phase participants were evaluated.
Time Frame: Baseline and Week 66
Population: mITT. Maintenance Phase Placebo/Placebo cohort is not reported since this is an exploratory population only. Results for the Induction phase populations for cohorts 1-3 are not presented
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 217 | 217
Percentage of Participants |  |  |  |  |  |  |  |  |  | 24.00 [18.77 to 30.06] | 35.00 [28.99 to 41.58]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.0088, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 11.3, 95% CI 2-sided [2.70 to 19.65] — Difference in response rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

6. Primary Outcome: Maintenance Phase: Percentage of Participants With Endoscopic Improvement at Week 66
Description: Endoscopic improvement is defined as 50% reduction from baseline in SES-CD score. Maintenance phase participants were evaluated.
Time Frame: Week 66
Population: mITT. Maintenance Phase Placebo/Placebo cohort is not reported since this is an exploratory population only. Induction Phase population for cohorts 1-3 are not included
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 217 | 217
Percentage of Participants |  |  |  |  |  |  |  |  |  | 12.2 [7.71 to 16.69] | 23.6 [17.90 to 29.29]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 11.5, 95% CI 2-sided [4.11 to 18.83] — Difference in response rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

7. Secondary Outcome: Induction Phase: Cohort 1: Percentage of Participants With Clinical Remission at Week 6
Description: Clinical remission is defined as SF mean daily score ≤3 and abdominal pain mean daily score ≤1, with no worsening in either subscore compared to baseline, averaged over the 7 days prior to visit.
Time Frame: Week 6
Population: mITT. Results for Induction Phase Cohort 2 and 3 and Maintenance Phase are not presented.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Groups:
- Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (210 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 5.1 [2.05 to 12.06] | 15.0 [10.41 to 21.13] | 24.8 [18.93 to 31.75] |  |  |  |  |  |  |  |

8. Secondary Outcome: Induction Phase: Cohort 2 and 3: Percentage of Participants With Clinical Remission at Week 6
Description: as for outcome 7
Time Frame: Week 6
Population: mITT. Results for Induction Phase Cohort 1 and Maintenance Phase are not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0
Percentage of Participants |  |  |  | 20.5 [15.16 to 27.01] | 21.3 [15.84 to 27.93] | 20.8 [13.91 to 30.00] | 23.8 [17.54 to 31.38] | 23.4 [17.29 to 30.97] |  |  |
Statistical Analysis 1: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 3.1, 95% CI 2-sided [-8.02 to 13.45] — Difference in remission rates are adjusted using CMH weights and the 95% CIs use the Newcombes method
Statistical Analysis 2: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Test type: Superiority; p = 0.7908, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 2.3, 95% CI 2-sided [-8.78 to 12.56] — Difference in remission rates are adjusted using CMH weights and the 95% CIs use the Newcombes method

9. Secondary Outcome: Induction Phase: Cohort 1: Percentage of Participants With SES-CD Score ≤4 (≤2 for Ileal Participants), With No Segment Having a Subcategory Score Greater Than (>)1, at Week 14
Description: Endoscopic Remission is defined as SES-CD total score <=4 (<=2 for ileal only patients), with no segment having a subcategory score >1. SES-CD = Simple Endoscopic Score for Crohn's Disease. A composite of four assessments, each rated from 0 to 3: size of ulcers, proportion of the surface covered by ulcers, proportion of the surface with any other lesions, and presence of narrowings (stenosis). The SES-CD total score ranges from 0 to 60, a higher score indicates worse disease activity.
Time Frame: Week 14
Population: mITT. Results for Induction Phase Cohort 2 and 3 and Maintenance Phase are not presented.
Measure: Number (90% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Percentage of Participants | 1.7 [-2.40 to 5.79] | 13.8 [7.53 to 20.14] | 8.3 [3.29 to 13.24] |  |  |  |  |  |  |  |

10. Secondary Outcome: Induction Phase: Cohort 2 and 3: Percentage of Participants With SES-CD Score ≤4 (≤2 for Ileal Participants), With No Segment Having a Subcategory Score Greater Than (>)1, at Week 14
Description: as for outcome 9
Time Frame: Week 14
Population: mITT. Results for Induction Phase Cohort 1 and Maintenance Phase are not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 176 | 174 | 96 | 143 | 145 | 0 | 0 | 0
Percentage of Participants |  |  |  | 9.9 [5.43 to 14.42] | 12.3 [5.43 to 14.42] | 8.7 [2.84 to 14.52] | 10.2 [5.15 to 15.27] | 15.3 [9.33 to 21.29] |  |  |
Statistical Analysis 1: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Test type: Superiority; p = 1, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 1.6, 95% CI 2-sided [-6.51 to 9.73] — Difference in remission rates are adjusted using CMH weights and the 95% CIs use the Newcombes method
Statistical Analysis 2: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Test type: Superiority; p = 0.5235, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 6.5, 95% CI 2-sided [-2.24 to 15.16] — Difference in remission rates are adjusted using CMH weights and the 95% CIs use the Newcombes method

11. Secondary Outcome: Induction Phase: Cohort 1: Change From Baseline in Crohn's Disease-Patient-Reported Outcome Signs and Symptoms (CD-PRO/SS) Score at Week 14
Description: CD-PRO/SS: Crohn's Disease Patient Reported Outcomes Signs and Symptoms. For each item, the score is taken as the average across 4-7 days eDiary data within a 9 day window from visit, else the score is considered missing. The CD-PRO/SS Bowel domain is a total score summed across 3 items and ranges from 0 - 16. The Functional domain score is a total score summed across 3 items and ranges from 0 - 12. A higher CD-PRO/SS score indicates worse quality of life. Participants are included in the analysis if they have both Baseline and at least one post-baseline score available.
Time Frame: Baseline and Week 14
Population: mITT. Data evaluable participants are included. Results for Induction Phase Cohort 2 and 3 and Maintenance Phase are not presented. Only patients with a baseline score and at least one post-baseline score are included in the analysis
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 46 | 76 | 87 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
scores on a scale
  CD-PRO/SS Functional Domain Score | -0.7 (0.4) | -1.4 (0.3) | -1.6 (0.3) |  |  |  |  |  |  |  |
  CD-PRO/SS Bowel Domain Score | -0.7 (0.4) | -1.5 (0.3) | -1.3 (0.3) |  |  |  |  |  |  |  |
Statistical Analysis 1: Comparison: Induction Phase - Cohort 1 (Exploratory): Placebo vs Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg; Bowel Domain Score; Test type: Superiority; p = 0.3110, MMRM; Difference in LSM = -0.5, 90% CI 2-sided [-1.4 to 0.3]

12. Secondary Outcome: Induction Phase: Cohort 2 and 3: Change From Baseline in Crohn's Disease-Patient-Reported Outcome Signs and Symptoms (CD-PRO/SS) Score at Week 14
Description: as for outcome 11
Time Frame: Baseline and Week 14
Population: mITT. Data evaluable participants are included. Results for Induction Phase Cohort 1 and Maintenance Phase are not presented. Only patients with a baseline score and at least one post-baseline score are included in the analysis
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 87 | 132 | 137 | 91 | 138 | 137 | 0 | 0 | 0
scores on a scale
  CD-PRO/SS Functional Domain Score: number analyzed (Participants) | 0 | 0 | 0 | 132 | 137 | 91 | 138 | 137 | 0 | 0 | 0
  CD-PRO/SS Functional Domain Score |  |  |  | -2.0 (0.2) | -2.3 (0.2) | -1.9 (0.3) | -1.6 (0.2) | -1.9 (0.2) |  |  |
  CD-PRO/SS Bowel Domain Score: number analyzed (Participants) | 0 | 0 | 0 | 132 | 137 | 91 | 138 | 137 | 0 | 0 | 0
  CD-PRO/SS Bowel Domain Score |  |  |  | -2.3 (0.3) | -2.2 (0.3) | -2.0 (0.3) | -2.0 (0.3) | -2.3 (0.3) |  |  |
Statistical Analysis 1: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Functional Domain Scale; Test type: Superiority; p = 1, MMRM — The multiplicity adjusted p-values are presented; Difference in LSM = 0.2, 95% CI 2-sided [-0.5 to 0.9]
Statistical Analysis 2: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Functional Domain Score; Test type: Superiority; p = 1, MMRM — The multiplicity adjusted p-values are presented; Difference in LSM = -0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 3: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg; Bowel Domain Score; Test type: Superiority; p = 1, MMRM — The multiplicity adjusted p-values are presented; Difference in LSM = 0.1, 95% CI 2-sided [-0.8 to 0.9]
Statistical Analysis 4: Comparison: Induction Phase - Cohort 3 (Pivotal): Placebo vs Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg; Bowel Domain Score; Test type: Superiority; p = 1, MMRM — The multiplicity adjusted p-values are presented; Difference in LSM = -0.3, 95% CI 2-sided [-1.1 to 0.5]

13. Secondary Outcome: Maintenance Phase: Percentage of Participants With Clinical Remission at Week 66, Among Those Who Achieved Clinical Remission at Week 14
Description: Clinical remission is defined as SF mean daily score ≤3 and abdominal pain mean daily score ≤1, with no worsening in either subscore compared to baseline, averaged over the 7 days prior to visit.
  Induction Phase Cohorts are not included
Time Frame: Baseline, Weeks 14 and 66
Population: mITT. Data evaluable participants are included. Placebo/Placebo Maintenance Cohort is not reported since this is an exploratory population only. Results for Induction Phase is not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 97 | 108
Percentage of Participants |  |  |  |  |  |  |  |  |  | 39.2 [30.05 to 49.12] | 56.5 [47.07 to 65.45]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.0677, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rate = 17.3, 95% CI 2-sided [3.52 to 30.27] — Difference in remission rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

14. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-Free Clinical Remission at Week 66, Among Those Who Were Receiving Corticosteroids at Baseline
Description: as for outcome 13
Time Frame: Baseline and Week 66
Population: mITT. Maintenance Phase Cohorts only. Placebo/Placebo Maintenance Cohort is not reported since this is an exploratory population only. Only patients receiving oral corticosteroids at Baseline are included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 91 | 93
Percentage of Participants |  |  |  |  |  |  |  |  |  | 11.0 [6.08 to 19.06] | 29.0 [20.79 to 38.94]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.0480, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rates = 18.6, 95% CI 2-sided [11.07 to 25.96] — Difference in remission rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

15. Secondary Outcome: Maintenance Phase: Percentage of Participants With Endoscopic Improvement at Week 66 Among Participants Who Achieved Endoscopic Improvement at Week 14
Description: Endoscopic improvement is defined as 50% reduction from baseline in SES-CD score. Induction Phase Cohorts are not included
Time Frame: Baseline, Weeks 14 and 66
Population: mITT. Only patients achieving endoscopic improvement at Week 14 are included in the analysis. Results for Induction Phase Cohort is not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 58 | 72
Percentage of Participants |  |  |  |  |  |  |  |  |  | 25.3 [14.14 to 36.44] | 37.5 [26.28 to 48.72]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.1210, Cochran-Mantel-Haenszel; Difference in rates = 13.5, 95% CI 2-sided [-2.90 to 29.94] — Difference in response rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

16. Secondary Outcome: Maintenance Phase: Percentage of Participants With SES-CD Score ≤4 (≤2 for Ileal Participants), With No Segment Having a Subcategory Score >1, at Week 66
Description: as for outcome 9
Time Frame: Week 66
Population: mITT. Maintenance Phase Placebo/Placebo are is not reported since this is an exploratory population only. Results for Induction Phase is not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 217 | 217
Percentage of Participants |  |  |  |  |  |  |  |  |  | 5.9 [2.62 to 9.18] | 12.1 [7.61 to 16.54]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.0480, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rates = 6.2, 95% CI 2-sided [0.54 to 11.93] — Difference in remission rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

17. Secondary Outcome: Maintenance Phase: Percentage of Participants With Durable Clinical Remission
Description: Clinical remission is defined as SF mean daily score ≤3 and abdominal pain mean daily score ≤1, with no worsening in either subscore compared to baseline, averaged over the 7 days prior to visit. Durable clinical remission was defined as clinical remission at ≥4 of the 6 in-clinic assessment visits conducted during the Maintenance Phase at Weeks 24, 28, 32, 44, 56, and 66. Induction Phase Cohorts are not included
Time Frame: Week 14 up to Week 66 (assessed at Weeks 24, 28, 32, 44, 56, and 66)
Population: mITT. Maintenance Phase Placebo/Placebo arm is not reported since this is an exploratory population only. Results for Induction Phase is not presented.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 217 | 217
Percentage of Participants |  |  |  |  |  |  |  |  |  | 19.8 [15.06 to 25.62] | 30.9 [25.11 to 37.31]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.0677, Cochran-Mantel-Haenszel — The multiplicity adjusted p-values are presented; Difference in rates = 11.2, 95% CI 2-sided [3.04 to 19.24] — Difference in response rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

18. Secondary Outcome: Maintenance Phase: Percentage of Participants With Corticosteroid-Free Clinical Remission for at Least 24 Weeks at Week 66, Among Those Who Were Receiving Corticosteroids at Baseline
Description: Clinical remission is defined as SF mean daily score ≤3 and abdominal pain mean daily score ≤1, with no worsening in either subscore compared to baseline, averaged over the 7 days prior to visit. Percentage of participants with clinical remission who will be off corticosteroids for at least 24 weeks prior to Week 66 will be reported.
  Induction Phase Cohorts are not included
Time Frame: Baseline and from Week 14 up to Week 66
Population: mITT. Maintenance Phase Placebo/Placebo is arm is not reported since this is an exploratory population only. Results for Induction Phase is not presented. Only patients receiving oral corticosteroids at Baseline are included in the analysis'
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 91 | 93
Percentage of Participants |  |  |  |  |  |  |  |  |  | 9.9 [5.29 to 17.74] | 25.8 [18.00 to 35.53]
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Test type: Superiority; p = 0.0035, Cochran-Mantel-Haenszel — Nominal p-value, no adjustment for multiplicity performed; Difference in rates = 16.2, 95% CI 2-sided [8.96 to 23.31] — Difference in remission rates is adjusted using CMH weights and the 95% CIs use the Newcombes method

19. Secondary Outcome: Maintenance Phase: Change From Baseline in CD-PRO/SS Score at Week 66
Description: as for outcome 11
Time Frame: Baseline and Week 66
Population: mITT. Data evaluable participants are included. Only patients with a baseline score and at least one post-baseline score are included in the analysis. The Maintenance Phase Placebo/Placebo arm is not reported since this is an exploratory population only. Results for Induction Phase is not presented.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 180 | 180
score on a scale
  Bowel |  |  |  |  |  |  |  |  |  | -1.7 (0.3) | -2.0 (0.3)
  Abdominal |  |  |  |  |  |  |  |  |  | -1.4 (0.2) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Functional Symptoms Domain; Test type: Superiority; p = 0.4009, MMRM — The multiplicity adjusted p-values are presented; Difference in LSM = -0.3, 95% CI 2-sided [-0.9 to 0.4]
Statistical Analysis 2: Comparison: Maintenance Phase - Etrolizumab Responders: Placebo vs Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg; Bowel Symptoms Domain; Test type: Superiority; p = 0.4009, MMRM — The multiplicity adjusted p-values are presented; Difference in LSM = -0.3, 95% CI 2-sided [-1.0 to 0.4]

20. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Adverse Event by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI-CTCAE v4.0)
Description: Investigator text for AEs is coded using MedDRA version 24.0. For participants counts, multiple occurrences of AEs in the same category for an individual are counted only once. For event counts, multiple occurrences of AEs in the same category for an individual are counted separately. Severity Grades from 1 to 5.
Time Frame: From Baseline up to Week 78
Population: Safety Population
Measure: Number; unit: Number of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217
Number of Participants | 50 | 83 | 82 | 120 | 115 | 51 | 95 | 85 | 42 | 190 | 189

21. Secondary Outcome: Overall Number of Participants With Adverse Events Leading to Study Drug Discontinuation
Description: Number of participants who discontinued the study due to the adverse events is reported.
Time Frame: From Baseline up to Week 78
Population: Safety Population
Measure: Number; unit: Number of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217
Number of Participants | 2 | 4 | 1 | 2 | 5 | 2 | 0 | 0 | 1 | 1 | 3

22. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Infection-Related Adverse Event by Severity, According to NCI-CTCAE v4.0
Description: Participants who Experienced at Least One Infection-Related Adverse Event by Severity, According to NCI-CTCAE v4.0 are reported. Grade 1 = mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; or intervention not indicated. Grade 2 = moderate; minimal, local, or non-invasive intervention indicated; or limiting age-appropriate instrumental activities of daily living. Grade 3 = severe or medically significant, but not immediately life-threatening; hospitalization indicated; disabling; or limiting self-care activities of daily living. Grade 4 = life-threatening consequences or urgent intervention indicated. Grade 5 = Death. The terms 'severe' and 'serious' are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs are counted only once per participant at the highest (worst) grade. Infections are identified by Primary System Organ Class term 'Infections and Infestations'
Time Frame: From Baseline up to Week 78
Population: Safety Population
Measure: Number; unit: Number of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217
Number of Participants
  Grade 1: number analyzed (Participants) | 11 | 30 | 32 | 66 | 50 | 16 | 40 | 42 | 22 | 121 | 106
  Grade 1 | 8 | 10 | 16 | 38 | 21 | 8 | 25 | 21 | 9 | 44 | 42
  Grade 2: number analyzed (Participants) | 11 | 30 | 32 | 66 | 50 | 16 | 40 | 42 | 22 | 121 | 106
  Grade 2 | 2 | 17 | 24 | 23 | 20 | 7 | 12 | 20 | 11 | 65 | 53
  Grade 3: number analyzed (Participants) | 11 | 30 | 32 | 66 | 50 | 16 | 40 | 42 | 22 | 121 | 106
  Grade 3 | 1 | 2 | 2 | 5 | 8 | 1 | 2 | 1 | 2 | 11 | 10
  Grade 4: number analyzed (Participants) | 11 | 30 | 32 | 66 | 50 | 16 | 40 | 42 | 22 | 121 | 106
  Grade 4 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
  Grade 5: number analyzed (Participants) | 11 | 30 | 32 | 66 | 50 | 16 | 40 | 42 | 22 | 121 | 106
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

23. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Infection-Related Serious Adverse Event
Description: Investigator text for AEs is coded using MedDRA version 24.0. Infections are identified by primary System Organ Class term 'Infections and Infestations'. The terms 'severe' and 'serious' are not synonymous and are independently assessed for each AE. Multiple occurrences of AEs in the same category for an individual are counted only once
Time Frame: From Baseline up to Week 78
Population: Safety Population
Measure: Number; unit: Number of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217
Number of Participants | 2 | 4 | 1 | 2 | 5 | 1 | 2 | 2 | 1 | 13 | 12

24. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Injection-Site Reaction by Severity, According to NCI-CTCAE v4.0
Description: Investigator test for AEs is coding using MedDRA version 24.0. Injection-Site Reactions are identified by eCRF checkbox for local injection site reactions, and/or primary or secondary HLT Injection Site Reactions. Multiple occurrences of AEs for an individual are counted only once, under the worst grade reported.
Time Frame: From Baseline up to Week 78
Population: Safety Population. Result data evaluable participants are included
Measure: Number; unit: Number of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217
Number of Participants
  Grade 1: number analyzed (Participants) | 4 | 7 | 4 | 10 | 9 | 1 | 11 | 6 | 3 | 18 | 9
  Grade 1 | 4 | 7 | 3 | 10 | 8 | 1 | 10 | 6 | 3 | 18 | 8
  Grade 2: number analyzed (Participants) | 4 | 7 | 4 | 10 | 9 | 1 | 11 | 6 | 3 | 18 | 9
  Grade 2 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1
  Grade 3: number analyzed (Participants) | 4 | 7 | 4 | 10 | 9 | 1 | 11 | 6 | 3 | 18 | 9
  Grade 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 4: number analyzed (Participants) | 4 | 7 | 4 | 10 | 9 | 1 | 11 | 6 | 3 | 18 | 9
  Grade 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 5: number analyzed (Participants) | 4 | 7 | 4 | 10 | 9 | 1 | 11 | 6 | 3 | 18 | 9
  Grade 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Overall Number of Participants Who Experienced at Least One Hypersensitivity Reaction by Severity, According to NCI-CTCAE v4.0
Description: Investigator text for AEs is coded using MedDRA version 24.0. Multiple occurrences of AEs for an individual are counted only once, under the worst grade reported.
Time Frame: From Baseline up to Week 78
Population: Safety Population. Result data evaluable participants are included
Measure: Number; unit: Number of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217
Number of Participants
  Grade 1: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 1 | 0 | 0 |  |  |  |  | 1 |  |  |  |
  Grade 2: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 2 | 2 | 1 |  |  |  |  | 0 |  |  |  |
  Grade 3: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 | 0 | 0 |  |  |  |  | 0 |  |  |  |
  Grade 4: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 4 | 0 | 0 |  |  |  |  | 0 |  |  |  |
  Grade 5: number analyzed (Participants) | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Grade 5 | 0 | 0 |  |  |  |  | 0 |  |  |  |

26. Secondary Outcome: Overall Number of Participants Who Develop Malignancies
Description: Participants with malignancies are reported. 'Malignancies are identified by SMQ Malignant and unspecified tumors (narrow)
Time Frame: From Baseline up to Week 78
Population: Safety Population
Measure: Number; unit: Number of Participants
Arm/Group | Induction Phase - Cohort 1 (Exploratory): Placebo | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 105 mg | Induction Phase - Cohort 1 (Exploratory): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 210 mg | Induction Phase - Cohort 2 (Open-Label): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Placebo | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 105 mg | Induction Phase - Cohort 3 (Pivotal): Etrolizumab 210 mg | Maintenance Phase - Placebo Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Placebo | Maintenance Phase - Etrolizumab Responders: Etrolizumab 105 mg
Number analyzed (Participants) | 59 | 120 | 121 | 176 | 174 | 96 | 143 | 145 | 53 | 217 | 217
Number of Participants | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1

27. Secondary Outcome: Percentage of Participants With Anti-Therapeutic Antibodies (ATAs) to Etrolizumab
Description: Participants who received at least one dose of study treatment and had at least one baseline or post-baseline ATA result. Induction: treatment groups were pooled across cohorts 1-3. Maintenance: treatment group is stratified by induction dose
Time Frame: Baseline, Pre-dose (Hour 0) on Weeks 4, 14, 24, 32, 44, 66 or early termination, 12 weeks after last dose (up to Week 78)
Population: Participants who received at least one dose of study treatment and had at least one baseline or post-baseline ATA result from at least one sample'. For the induction phase, participants for cohorts 1-3 were pooled across each dose arm. For maintenance phase, participants were grouped according to their induction & maintenance treatment arms
Measure: Number; unit: Percentage of Participants
Groups:
- Etro 105mg Induction Only Cohort: Etro 105mg Induction Only Cohort Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8 and 12
- Etro 210mg Induction Only Cohort: Induction only cohort. Participants randomized to this arm received one SC injection of etrolizumab (210 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8 and 12
- Etro 105/ Placebo Induction and Maintenance Phase Cohort: Etro 105/ Placebo Induction and Maintenance Phase Cohort
  Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy that were re-randomized into the Mainetnance Phase. Etrolizumab responders from induction who re re-randomized to this arm received blinded maintenance treatment with an SC injection of placebo q4w from Week 16 to Week 64
- Etro 210/ Placebo Induction and Maintenance Phase: Participants who received etrolizumab 210 mg during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy that were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who were re-randomized to this arm received blinded maintenance treatment with an SC injection of placebo q4w from Week 16 to Week 64
- Etro 105/Etro 105 Induction and Maintenance Phase: Participants who received etrolizumab 105mg during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy that were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who were re-randomized to this arm received blinded maintenance treatment with an SC injection of etrolizumab 105mg q4w from Week 16 to Week 64
- Etro 210/Etro 105 Induction and Maintenance Phase: Participants who received etrolizumab 210mg during the Induction Phase (from Cohorts 1-3) and achieved CDAI-70 response at Week 14 without the use of rescue therapy that were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who were re-randomized to this arm received blinded maintenance treatment with an SC injection of etrolizumab 105mg q4w from Week 16 to Week 64
Arm/Group | Etro 105mg Induction Only Cohort | Etro 210mg Induction Only Cohort | Etro 105/ Placebo Induction and Maintenance Phase Cohort | Etro 210/ Placebo Induction and Maintenance Phase | Etro 105/Etro 105 Induction and Maintenance Phase | Etro 210/Etro 105 Induction and Maintenance Phase
Number analyzed (Participants) | 222 | 223 | 108 | 109 | 109 | 108
Percentage of Participants
  Baseline with positive ADA: number analyzed (Participants) | 217 | 218 | 107 | 108 | 107 | 108
  Baseline with positive ADA | 4.1 | 2.8 | 2.8 | 5.6 | 2.8 | 0
  Treatment emergent ADA: number analyzed (Participants) | 213 | 216 | 108 | 109 | 109 | 108
  Treatment emergent ADA | 23 | 22.7 | 23.1 | 33.9 | 33.9 | 21.3

28. Secondary Outcome: Observed Trough Serum Concentration (Ctrough) of Etrolizumab
Description: Serum Etrolizumab Trough Concentration
Time Frame: Induction Phase at Weeks 10 and 14, Maintenance Phase at Weeks 16, 24, 28, 32, 44, and 66
Population: mITT. All participants who received at least one dose of study drug and had evaluable PK data
Measure: Mean (Standard Deviation); unit: microgram/mL
Groups:
- Cohort 1 Etrolizumab 105mg: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Cohort 1 Etrolizumab 210mg: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one subcutaneous (SC) injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Cohort 2 Etrolizumab 105mg: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking of the dose of etrolizumab, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Cohort 2 Etrolizumab 210mg: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking for the dose of etrolizumab, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Cohort 3 Etrolizumab 105mg: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (105 mg) at Weeks 0, 4, 8, 12 and one SC injection of etrolizumab-matching placebo at Week 2 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Cohort 3 Etrolizumab 210mg: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Maintenance Phase - Etrolizumab 105 mg/ Etrolizumab 105 mg: Participants who received etrolizumab 105 mg during Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response without the use of resceu therapy will be re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm will receive blinded maintenance treatment with an SC injection of etrolizumab 105 mg q4w from Week 16 to Week 64
- Maintenance Phase - Etrolizumab 210 mg/ Etrolizumab 105 mg: Participants who received etrolizumab 210 mg during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy will be re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm will receive blinded maintenance treatment with an SC injection of etrolizumab (105 mg) q4w from Week 16 to Week 64.
Arm/Group | Cohort 1 Etrolizumab 105mg | Cohort 1 Etrolizumab 210mg | Cohort 2 Etrolizumab 105mg | Cohort 2 Etrolizumab 210mg | Cohort 3 Etrolizumab 105mg | Cohort 3 Etrolizumab 210mg | Maintenance Phase - Etrolizumab 105 mg/ Etrolizumab 105 mg | Maintenance Phase - Etrolizumab 210 mg/ Etrolizumab 105 mg
Number analyzed (Participants) | 117 | 121 | 175 | 172 | 138 | 141 | 109 | 108
microgram/mL
  Week 10: number analyzed (Participants) | 104 | 112 | 158 | 160 | 124 | 126 | 0 | 0
  Week 10 | 9.39 (4.59) | 25.1 (11.6) | 10.3 (5.07) | 25.7 (11.9) | 9.78 (4.63) | 25.5 (11.0) |  |
  Week 14: number analyzed (Participants) | 96 | 103 | 148 | 144 | 115 | 120 | 0 | 0
  Week 14 | 10.2 (5.27) | 23.2 (10.6) | 11.0 (5.04) | 24.1 (11.4) | 10.8 (5.43) | 24.6 (9.53) |  |
  Week 16: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 102 | 94
  Week 16 |  |  |  |  |  |  | 6.15 (4.20) | 14.8 (10.5)
  Week 24: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 96 | 97
  Week 24 |  |  |  |  |  |  | 6.58 (4.59) | 8.20 (6.34)
  Week 28: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 88 | 82
  Week 28 |  |  |  |  |  |  | 7.29 (8.45) | 8.07 (5.81)
  Week 32: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 85 | 81
  Week 32 |  |  |  |  |  |  | 7.13 (9.76) | 7.89 (5.96)
  Week 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 68 | 73
  Week 44 |  |  |  |  |  |  | 6.68 (3.75) | 8.31 (6.68)
  Week 66: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 61 | 63
  Week 66 |  |  |  |  |  |  | 11.7 (5.82) | 12.2 (6.44)

ADVERSE EVENTS:
Time Frame: From Baseline up to a maximum of 78 weeks
Groups:
- Etrolizumab 210mg Cohort 1: Cohort 1 enrolled participants first before Cohorts 2 and 3 in order to conduct an exploratory analysis on induction data. Participants randomized to this arm received one subcutaneous (SC) injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Etrolizumab 210mg Cohort 2: Cohort 2 enrolled participants after Cohort 1 and was considered a "feeder" cohort to help achieve the necessary sample size for the Maintenance Phase. Participants randomized to this arm received one SC injection of open-label etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking for the dose of etrolizumab, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Etrolizumab 210mg Cohort 3: Cohort 3 was the last to enroll participants (after Cohort 2) and was the pivotal cohort for the Induction Phase. Participants randomized to this arm received one SC injection of etrolizumab (210 mg) at Weeks 0, 2, 4, 8, and 12 during the 14-week Induction Phase. In order to preserve the masking, participants also received one SC injection of etrolizumab-matching placebo at Weeks 0, 4, 8, and 12.
- Etrolizumab/Placebo: Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm received blinded maintenance treatment with an SC injection of placebo q4w from Week 16 to Week 64.
- Etrolizumab/Etrolizumab 105mg: Participants who received etrolizumab during the Induction Phase (from Cohorts 1-3) and achieved a CDAI-70 response at Week 14 without the use of rescue therapy were re-randomized into the Maintenance Phase. Etrolizumab responders from induction who are re-randomized to this arm received blinded maintenance treatment with an SC injection of etrolizumab (105 mg) q4w from Week 16 to Week 64.
Arm/Group | Placebo Cohort 1 | Etrolizumab 105mg Cohort 1 | Etrolizumab 210mg Cohort 1 | Etrolizumab 105mg Cohort 2 | Etrolizumab 210mg Cohort 2 | Placebo Cohort 3 | Etrolizumab 105mg Cohort 3 | Etrolizumab 210mg Cohort 3 | Placebo/Placebo | Etrolizumab/Placebo | Etrolizumab/Etrolizumab 105mg
All-Cause Mortality (participants affected / at risk) | 0/59 | 0/120 | 0/121 | 0/176 | 0/174 | 0/96 | 0/143 | 0/145 | 0/53 | 0/217 | 1/217
Serious Adverse Events (participants affected / at risk) | 8/59 | 20/120 | 12/121 | 18/176 | 20/174 | 8/96 | 12/143 | 8/145 | 9/53 | 33/217 | 30/217
Other Adverse Events (participants affected / at risk) | 32/59 | 61/120 | 52/121 | 80/176 | 68/174 | 35/96 | 65/143 | 45/145 | 33/53 | 154/217 | 147/217
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort 1 (N=59) | Etrolizumab 105mg Cohort 1 (N=120) | Etrolizumab 210mg Cohort 1 (N=121) | Etrolizumab 105mg Cohort 2 (N=176) | Etrolizumab 210mg Cohort 2 (N=174) | Placebo Cohort 3 (N=96) | Etrolizumab 105mg Cohort 3 (N=143) | Etrolizumab 210mg Cohort 3 (N=145) | Placebo/Placebo (N=53) | Etrolizumab/Placebo (N=217) | Etrolizumab/Etrolizumab 105mg (N=217)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Crohn's disease (Gastrointestinal disorders) | 6 (9) | 12 (12) | 7 (7) | 5 (6) | 10 (11) | 3 (3) | 7 (8) | 5 (5) | 4 (4) | 14 (15) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Optic neuropathy (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Granuloma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess intestinal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis listeria (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral gas embolism (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Removal of foreign body from gastrointestinal tract (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Cohort 1 (N=59) | Etrolizumab 105mg Cohort 1 (N=120) | Etrolizumab 210mg Cohort 1 (N=121) | Etrolizumab 105mg Cohort 2 (N=176) | Etrolizumab 210mg Cohort 2 (N=174) | Placebo Cohort 3 (N=96) | Etrolizumab 105mg Cohort 3 (N=143) | Etrolizumab 210mg Cohort 3 (N=145) | Placebo/Placebo (N=53) | Etrolizumab/Placebo (N=217) | Etrolizumab/Etrolizumab 105mg (N=217)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 5 (5) | 2 (2) | 5 (5) | 4 (4) | 2 (2) | 10 (11) | 11 (12)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (7) | 10 (12) | 14 (16) | 10 (16) | 13 (15) | 10 (11) | 6 (6) | 9 (12) | 24 (29) | 27 (34)
Crohn's disease (Gastrointestinal disorders) | 12 (14) | 9 (12) | 8 (9) | 13 (13) | 7 (7) | 3 (3) | 7 (8) | 8 (9) | 13 (13) | 63 (66) | 37 (43)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 6 (7) | 2 (2) | 12 (15) | 21 (22)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 5 (5) | 0 (0) | 4 (4) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 11 (11) | 8 (8)
Frequent bowel movements (Gastrointestinal disorders) | 1 (2) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 7 (8) | 8 (14) | 6 (6) | 11 (14) | 8 (11) | 6 (6) | 6 (7) | 3 (7) | 13 (16) | 21 (28)
Vomiting (Gastrointestinal disorders) | 2 (2) | 7 (9) | 6 (8) | 4 (5) | 3 (3) | 2 (3) | 4 (4) | 4 (4) | 0 (0) | 12 (22) | 14 (16)
Fatigue (General disorders) | 1 (1) | 4 (4) | 3 (3) | 6 (7) | 2 (2) | 3 (5) | 4 (5) | 5 (6) | 1 (1) | 10 (11) | 13 (15)
Injection site erythema (General disorders) | 3 (5) | 5 (12) | 3 (7) | 9 (18) | 7 (14) | 0 (0) | 6 (8) | 5 (9) | 2 (4) | 14 (41) | 7 (16)
Pyrexia (General disorders) | 0 (0) | 4 (4) | 4 (4) | 5 (5) | 5 (5) | 2 (2) | 6 (8) | 4 (4) | 3 (3) | 16 (18) | 7 (7)
Influenza (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 7 (7) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 15 (16) | 6 (6)
Nasopharyngitis (Infections and infestations) | 2 (2) | 7 (7) | 9 (13) | 11 (12) | 7 (7) | 4 (4) | 7 (9) | 9 (9) | 3 (3) | 27 (35) | 32 (42)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 6 (9) | 13 (16)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 6 (6) | 1 (1) | 11 (13) | 7 (7) | 1 (1) | 5 (5) | 4 (6) | 3 (3) | 26 (30) | 16 (19)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 6 (7) | 8 (9) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 13 (13) | 11 (18)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (6) | 10 (10) | 12 (13) | 9 (11) | 7 (7) | 11 (12) | 7 (8) | 9 (12) | 25 (30) | 27 (32)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 4 (4) | 4 (4) | 1 (1) | 3 (3) | 2 (2) | 0 (0) | 5 (5) | 10 (10) | 4 (5)
Headache (Nervous system disorders) | 4 (5) | 13 (14) | 7 (10) | 20 (27) | 20 (22) | 7 (10) | 14 (20) | 8 (15) | 4 (4) | 27 (43) | 22 (27)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 3 (3) | 4 (5) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/28/NCT02394028/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT02394028/SAP_001.pdf